CLINICAL TRIAL: NCT04531501
Title: COVID-19 Saliva Test Research Study - Evaluation of High Throughput COVID-19 Testing Via Saliva Based Sampling and Alternative RNA Extraction Methods.
Brief Title: COVID-19 Saliva Test Research Study
Status: Completed | Type: Observational
Sponsor: Chronomics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 283560
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Patients suspected to have Covid-19: Individuals suspected to have COVID-19 who are admitted to Gloucestershire Hospitals NHS Foundation Trust facilities for treatment for COVID-19. Individuals with full mental capacity.
  Interventions: Diagnostic Test: Saliva and NPS test
- Patients tested positive for Covid-19: Individuals tested positive for COVID-19 at Northern Care Alliance NHS Group using an NHS NPS test who are accessible within 24 hours and consent to providing a saliva sample and further NPS sample for Chronomics.
  Interventions: Diagnostic Test: Saliva and NPS test

INTERVENTIONS:
Diagnostic Test: Saliva and NPS test — N/A Our study will not impact their path of care as they will be doing an NHS test which will determine their path of care at the NHS

SUMMARY:
The objective of this study is to compare the Chronomics test against the NPS tests and protocol currently in use to demonstrate the efficacy of Chronomics' approach. The principal question is: Does the Chronomics saliva based test perform as well as the NPS NHS test?

DETAILED DESCRIPTION:
In December 2019, a novel coronavirus caused an outbreak in Wuhan, China. Just a month later, Covid-19 was declared a Public Health Emergency of International Concern on 30 January 2020. The World Health Organisation (WHO) repeatedly announced that 'Diagnostic testing for COVID-19 is critical to tracking the virus, understanding epidemiology, informing case management, and to suppressing transmission'. The priority within Public Health England (PHE) was to scale up public health testing using molecular diagnosis through real-time RT-PCR (RdRp gene) assay based on oral swabs.

Some of the key challenges publicly presented regarding testing are speed of mobilisation, supply chain issues due to the international demand for crucial testing materials like kits, swabs and chemical reagents, and the quality and comfort of the nasopharyngeal (NSP) swabs commonly used.

Chronomics has developed novel methods to address these problems. Firstly, due to the shortage of the specific branded reagent products used in the official CDC FDA EUA COVID-19 RT-qPCR protocol for RNA extraction, Chronomics have sourced and compiled testing of components to create an extraction kit with greater availability of supply for use within the protocol. Secondly, Chronomics' methods are based on saliva collection which are pain-free and easy to collect.

The objective of this study is to compare the Chronomics test against the NPS tests and protocol currently in use to demonstrate the efficacy of Chronomics' approach. The principal question is: Does the Chronomics saliva based test perform as well as the NPS NHS test? There are two components of Chronomics' testing framework that the investigators are looking to validate to feed into this. Firstly, that Chronomics' alternative reagents and workflow (RNA-extraction and RT-PCR steps) do not impact sensitivity of detection and secondly, that Chronomics' alternative sampling source of saliva also does not impact sensitivity of detection. To achieve validation of these two components, the investigators will compare both a Chronomics saliva sample vs an NHS NPS sample, and a Chronomics NPS sample vs an NHS NPS sample. The investigators would require access to the output (and information as to the linked patient) for the NHS gold-standard workflow.

ELIGIBILITY:
Site 1: Testing on Admission approach Inclusion Criteria Individuals suspected to have COVID-19 who were admitted to Gloucestershire Hospitals NHS Foundation Trust facilities for treatment for COVID-19. Individuals with full mental capacity.

Exclusion Criteria None

Site 2: Positive Matching approach Inclusion Criteria Individuals tested positive for COVID-19 at Northern Care Alliance NHS Group using an NHS NPS test who are accessible within 24 hours and consent to providing a saliva sample and further NPS sample for Chronomics.

Exclusion Criteria Individuals who have not tested at all or have not tested positive.

Ages: 18 Years to 117 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study is being conducted at specific hospitals so will apply geographically to people within the eligibility criteria as described above.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Test Result | Within 2 weeks of sample collection
  Positive / Negative / Indeterminate

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Gloucestershire Royal Hospital, Gloucester
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No